CLINICAL TRIAL: NCT02651051
Title: The Influence of Whey Protein Addition to a Fat-based Breakfast on Metabolic and Appetite Parameters Following a Second Meal
Brief Title: Metabolic and Appetite Parameters Following Addition of Whey Protein to a Fat-based Breakfast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HLS-13-131017b
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Postprandial glycemia; Metabolic health measures
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Fat Breakfast Meal (Sham Comparator): High fat breakfast meal served without addition of whey protein isolate
  Interventions: Other: High Fat Breakfast Meal
- High Fat Breakfast Meal + Whey Protein (Experimental): High fat breakfast meal served with addition of whey protein isolate
  Interventions: Dietary Supplement: Whey Protein; Other: High Fat Breakfast Meal

INTERVENTIONS:
Dietary Supplement: Whey Protein — 20 g whey protein isolate (Arla Foods Ingredients Group) added to breakfast meal
  Arms: High Fat Breakfast Meal + Whey Protein
Other: High Fat Breakfast Meal — A standardised high fat breakfast served to all participants. The macronutrient distribution of the breakfast is 12% protein, 3% carbohydrate, 85% fat (1771 kJ; 423 kcal total)

SUMMARY:
The purpose of this study is to investigate whether the addition of whey protein to a breakfast high in fat content will influence acute metabolic and appetite responses, as well as responses to a subsequent lunch meal.

DETAILED DESCRIPTION:
Participants will be asked to report to the lab for their first main trial, having not eaten for 12 hours, and refrained from caffeine and alcohol intake and strenuous exercise for 24 hours. Both trials will take place at the same time of day.

Upon arrival height and body mass will be recorded and a cannula will be inserted into a vein in the back of the hand and a 10 ml blood sample will be taken.A visual analogue scale (VAS) will then be used to subjectively measure the participant's appetite pre-breakfast.

Participants will then be provided with one of the two breakfast meals that are being tested in a randomised order. The two breakfasts consist of a high fat breakfast or high fat plus additional whey protein. A drink of water shall also be consumed, the volume of which depends on the trial being carried out. The high fat breakfast will consist of scrambled egg yolks made with single cream and butter (Tesco, Hertfordshire, UK). The macronutrient distribution of the breakfast is 12% protein, 3% carbohydrate, 85% fat (1771 kJ; 423 kcal total). For the whey protein trial, 23.9g whey protein isolate (Lacprodan DI-9224, Arla Foods, Denmark) shall be added to water and incorporated into each meal as a drink on the side, in order to provide 20g whey protein.

A timer shall be set when the participant takes their first mouthful of breakfast, and they will be required to rest for the following 3 hours. At 15, 30, 45, 60, 90, 120, 150 and 180 minutes post-breakfast 10 ml blood samples shall be collected. Every 30 minutes during this period the appetite VAS will also be completed. After this participants will be provided with a standardised lunch meal which shall consist of pasta with a tomato and basil sauce, olive oil and cheddar cheese, along with a 350 ml drink of water. The macronutrient distribution of the lunch is 13% protein, 49% carbohydrate, 38% fat. Following this, the post-breakfast procedure shall be repeated for another period of 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 years old (male)
* Recreationally active (>30 minutes of structured exercise, 5 times/week)

Exclusion Criteria:

* Metabolic disease (e.g. Type 2 diabetes, thyroid disorders)
* Taking any prescribed medication
* Regular breakfast skipper
* Food allergies or intolerances
* Eating disorders
* Smoker

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose responses | 0-360 minutes post breakfast
  Blood glucose concentration determined in whole blood sampled at regular intervals post-breakfast and post-lunch

SECONDARY OUTCOMES:
Acute subjective appetite responses | 0-360 minutes post breakfast
  Subjective appetite ratings determined from Visual Analogue Scales sampled at regular intervals

CONTACTS AND LOCATIONS:
Overall Officials: Emma J Stevenson, PhD, Study Director — Northumbria University
Locations (1):
- Faculty of Health and Life Sciences, Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom